CLINICAL TRIAL: NCT01067339
Title: Lp-PLA2, Progenitor Cells and Coronary Atherosclerosis in Humans AIM III
Brief Title: Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Progenitor Cells and Coronary Atherosclerosis in Humans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GlaxoSmithKline (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amir Lerman, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-000044; 5R01HL092954 (NIH); 5R01AG031750 (NIH)
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Endothelial Dysfunction
Keywords: coronary endothelial dysfunction; coronary vasospasm
MeSH Terms: conditions — Coronary Vasospasm | interventions — darapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darapladib (Experimental): Subjects randomized to this arm will receive a darapladib tablet, 160 mg, by mouth, once per day for 6 months.
  Interventions: Drug: darapladib
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive a placebo tablet matching the study drug, once per day for 6 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: darapladib — darapladib, tablet, 160 mg, by mouth, one time daily, 6 month duration
  Arms: Darapladib
Drug: placebo — placebo, by mouth, once daily for six months
  Arms: Placebo

SUMMARY:
AIM III is a prospective, randomized, double-blinded, placebo controlled trial. The study is directly connected to IRB 08-008161 as a specific aim of the National Institute of Health (NIH) grant. Participants may either consent to and qualify for AIM I and AIM II (IRB 08-008161) or have a cardiac catheterization with acetylcholine testing in the Cardiac Catheterization Laboratory at Mayo Clinic in Rochester, Minnesota to be considered for this study.

DETAILED DESCRIPTION:
The main goal of AIM III is to assess and quantify the effect of long-term administration of darapladib 160 mg once a day, a selective, reversible, orally active inhibitor of plasma and vascular Lp-PLA2, on coronary endothelial function, progression of coronary atherosclerosis as determined by intravascular ultrasound (IVUS), and atherosclerosis in patients with early atherosclerosis. Patients with evidence of coronary endothelial dysfunction, as determined by intracoronary administration of acetylcholine during angiography and IVUS, will be followed for 6 months during once daily dosing of darapladib. Coronary endothelial function is determined by the changes in coronary artery diameter and coronary blood flow response to the intracoronary administration of acetylcholine and adenosine. The patients will be followed in clinic 6 months. They will have follow-up angiography, assessment of endothelial function, and IVUS during the six month visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing coronary angiography including endothelial function testing with the medication acetylcholine in the cardiac catheterization laboratory at Mayo Clinic. Patients may be enrolled in AIM I and AIM II IRB 08-008161 :Lp-PLA2, Progenitor Cells and Atherosclerosis in Humans".
2. Male or female aged at least 18 years, inclusive, at screening. Female subjects must be post-menopausal or using a highly effective method for avoidance of pregnancy. The decision to include or exclude women of childbearing potential may be made at the discretion of the investigator in accordance with local practice in relation to adequate contraception.
3. Age greater than 18 up to age 85

Exclusion Criteria:

1. Current severe heart failure New York Heart Association class III or IV with ejection fraction less than 40%
2. Unstable angina
3. Myocardial infarction or angioplasty within 6 months prior to entry into the study
4. Planned coronary revascularization (PCI or CABG)
5. Planned major surgical procedure
6. Patients with segments with endothelial dysfunction of less than 10 mm in length or complete occlusion will be excluded.
7. Angiographic exclusion criteria include left main disease with greater than 30% stenosis on angiogram, luminal diameter of the study vessel less than 2.5 mm, severe tortuousity of the study vessel, or any other relevant anatomical reasons that the investigator deems inappropriate for the study.
8. Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence of abnormal liver function tests (total bilirubin or alkaline phosphatase > 1.5 x upper limit of normal (UNL); or alanine transaminase (ALT) or aspartate amino transferase (AST) > 2.5 x UNL or other hepatic abnormalities that in the opinion of the investigator would preclude the subject from participation in the study.
9. Chronic or acute kidney disease with serum creatinine greater than or equal to 2 mg/dL or estimated glomerular filtration rate <40 mL/min/1.73m2, renal transplant status, history of contrast nephropathy,
10. Poorly controlled hypertension despite lifestyle modifications and pharmacotherapy. (systolic BP >160 mm Hg and/or diastolic BP >110 mm Hg),
11. Poorly controlled diabetes mellitus (HbA1c >10%),
12. Current or within 1 month use of any form of corticosteroids,
13. Severe asthma that is poorly controlled on pharmacotherapy
14. History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions
15. Current life-threatening conditions other than vascular disease, alcohol or drug abuse within the last 6 months
16. Malignancy within the past 5 years,
17. Positive pregnancy test (all female subjects of childbearing potential must have a urine β-human chorionic gonadotropin (hCG) pregnancy test performed at Screening and/or within 7 days prior to randomization) or is known to be pregnant or lactating.
18. Current or planned chronic administration of strong oral or injectable cytochrome P-450 isoenzyme 3A4 (CYP3A4) inhibitors.
19. Subjects with both parents of Japanese, Chinese, or Korean ancestry must have a blood sample collected for assessment of Lp-PLA2 activity by the central laboratory prior to randomization. Those with Lp-PLA2 activity ≤10 nmol/min/mL will be excluded from participation in the study.
20. Previous exposure to darapladib (SB-480848).
21. Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of the study medication, or any subject the investigator deems unsuitable for the study
22. Patients who require treatment with positive inotropic agents other than digoxin during the study
23. Patients with cerebrovascular accident within 6 months prior to entry into the study
24. Significant endocrine, hepatic or renal disorders
25. Local or systemic infectious disease within 4 weeks prior to entry into study
26. Mental instability
27. Federal Medical Center inmates
28. Hemoglobin less than 12 mg/dL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-02-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prasad M, Lennon R, Barsness GW, Prasad A, Gulati R, Lerman LO, Lerman A. Chronic inhibition of lipoprotein-associated phospholipase A2 does not improve coronary endothelial function: A prospective, randomized-controlled trial. Int J Cardiol. 2018 Feb 15;253:7-13. doi: 10.1016/j.ijcard.2017.09.171. PMID 29306475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic in Rochester, Minnesota between February 2010 and February 2015.
Pre-assignment Details: 70 subjects signed informed consent, but 5 subjects withdrew (subject decision) prior to randomization.
Period: Overall Study
Arm/Group | Darapladib | Placebo
Started | 31 | 34
Completed | 25 | 29
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Population: The baseline characteristics table only includes subjects who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Darapladib | Placebo | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.7) | 54.0 (10.5) | 54.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 26 | 43
  Male | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Coronary Artery Diameter
Description: The change of coronary artery diameter was measured in response to a maximal dose of acetylcholine administered intracoronary during an invasive coronary endothelial function assessment. Percentage change in coronary artery diameter provides a measure of endothelium dependent epicardial function.
Time Frame: baseline, six months
Measure: Mean (Inter-Quartile Range); unit: % change coronary artery diameter
Arm/Group | Darapladib | Placebo
Number analyzed (Participants) | 25 | 29
% change coronary artery diameter | 3 [-9 to 15] | 3 [-12 to 19]

2. Primary Outcome: Percentage Change in Coronary Blood Flow (CBF)
Description: The change in coronary blood flow was measured in response to maximal dose of acetylcholine administered intracoronary during an invasive coronary endothelial function assessment. Percentage change in coronary blood flow provides a measure of endothelium dependent microvascular function.
Time Frame: baseline, six months
Measure: Mean (Inter-Quartile Range); unit: % change coronary blood flow
Arm/Group | Darapladib | Placebo
Number analyzed (Participants) | 25 | 29
% change coronary blood flow | -5 [-24 to 54] | 39 [-26 to 67]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Darapladib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/34
Serious Adverse Events (participants affected / at risk) | 2/31 | 3/34
Other Adverse Events (participants affected / at risk) | 6/31 | 16/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darapladib (N=31) | Placebo (N=34)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) — Reported to ER due to chest pain not relieved with sub-lingual nitroglycerin.
Hematoma in groin (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darapladib (N=31) | Placebo (N=34)
Cough, chest congestion, viral (Infections and infestations) | 0 (0) | 1 (1)
Fluid retention (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 2 (2) | 1 (1)
Overdose (Surgical and medical procedures) | 0 (0) | 1 (1) — Overdose on sedative hypnotic Hospitalized for 5 days. This even occured prior to subject starting study medication/placebo.
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin abcess on abdomen
Oral Thrush (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Lower extremity edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Scalp laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — scalp laceration requiring 3 staples secondary to a fall while working in barn
Fracture right wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Irregular heart rate (Cardiac disorders) | 0 (0) | 1 (1)
Sweating around torso about 2 hours after taking study medication (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Product Issues) | 0 (0) | 1 (1) — Allergic reaction, facial swelling and rash. Suspect Norvasc. Subject stopped Norvasc.
Hypotension (Product Issues) | 0 (0) | 1 (1) — Hypotension: Subject notes episodes of hypotension to 75/40. She relates a lower blood pressure to ingestion of L-Arginine.
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Diverticulitis with cramping and frequent diarrhea.
Diarrhea (Product Issues) | 0 (0) | 1 (1) — Diarrhea lasting 2 days. Patient states this started after she took Mucinex. It resolved when she stopped the medication.
Bone spur (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Bone spur right ankle noted after developing pain in the area. Surgical removal of the bone spur following completion of the study.
Chest discomfort/angina (Cardiac disorders) | 3 (3) | 1 (1)
Vaginal yeast infection (Infections and infestations) | 0 (0) | 2 (2)
Abdominal cramping and diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Abdominal cramping and diarrhea. Held L-Arginine for several days. Noted partial resolution.
Muscle aches (Product Issues) | 0 (0) | 1 (1) — Noting muscle aching in the long muscles of the legs at night. Taking Crestor 40 mg daily. Reduced Crestor dose.
Inpatient psychiatric admission for pre-existing biolar disorder. (Nervous system disorders) | 0 (0) | 1 (1)
Myocardial bridge (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) — Chest pain. Ruled out cardiac cause.
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Fibromyalgia with significant muscle spasm.
Difficulty swallowing medications (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — back pain related to fall on ice.
Anomalous pulmonary vein and tricuspid valve repair (Cardiac disorders) | 1 (1) | 0 (0) — Hospitalization for repair of anomalous pulmonary vein and tricuspid valve repair. Both diagnosis known prior to study start. Surgery planned for after study but changed due to increasing severity of chest pain. No significant complications.
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes